CLINICAL TRIAL: NCT02729545
Title: The Efficacy and Safety Study of Tung's Acupuncture for Improving Ovarian Function of Polycystic Ovarian Syndrome: a Randomised Controlled Trial
Brief Title: The Efficacy and Safety Study of Tung's Acupuncture for Polycystic Ovarian Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JJ2015-42
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: acupuncture; LH/FSH; total testosterone (TT); polycystic ovarian syndrome(PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Cyproterone Acetate; Ethinyl Estradiol; Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Intervention Model Description: The study was a randomized, drug-controlled, and parallel group trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tung's acupuncture (Experimental): The Tung's acupuncture group received acupuncture treatments twice per week for 12 weeks. The study took Tung's acupoints as main acupuncture points, which were Fuke, Huanchao, Tianhuang, Renhuang, as well as the traditional acupoints Guanyuan (CV4) and Zigong (EX-CA1).
  Interventions: Other: Tung's acupuncture
- CPA/EE (Active Comparator): Cyproterone acetate/ethinylestradiol (CPA/EE) was taken orally one tablet per day from the 8th day of menstrual cycle or any day for patients with amenorrhea. The pills were administered for 21 days consecutively. The patients then stopped taking the pills for seven days and, on the eighth day, continued to take the pills again for three menstrual cycles (28 day cycles).
  Interventions: Drug: Cyproterone acetate/ethinylestradiol (CPA/EE)

INTERVENTIONS:
Other: Tung's acupuncture — The study took Tung's acupoints as main acupuncture points, which were Fuke, Huanchao, Tianhuang, Renhuang, as well as the traditional acupoints Guanyuan (CV4) and Zigong (EX-CA1).
  Arms: Tung's acupuncture
Drug: Cyproterone acetate/ethinylestradiol (CPA/EE) — Cyproterone acetate/ethinylestradiol (CPA/EE) contains 2mg cyproterone acetate (an anti-androgenic progestin) and 0.035mg ethinylestradiol (CPA/EE). The pills were administered for 21 days consecutively. The patients then stopped taking the pills for seven days and, on the eighth day, continued to take the pills again for three menstrual cycles (28 day cycles).
  Other Names: Diane-35
  Arms: CPA/EE

SUMMARY:
This study evaluates the efficacy and safety in improving ovarian function of polycystic ovarian syndrome in adults. Half of patients will receive Tung's acupuncture therapy, while the other half will receive Diane-35(CPA/EE) as the control group.

DETAILED DESCRIPTION:
Both Tung's acupuncture therapy and Diane-35(CPA/EE) could improve the symptom of patients with polycystic ovarian syndrome, but until now there is no definite evidence to indicate acupuncture could play the same role in improving ovarian function. So we design this study to observe the change of follicular development, ovary size and sex hormone( testosterone, follitropin, luteinizing hormone) before and after the treatment, and evaluate the efficacy and safty of acupuncture.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese;
2. 18-45 years old;
3. to meet the diagnostic criteria for polycystic ovary syndrome;
4. no need for pregnancy in the next six months;
5. volunteering to join this research and give informed consent prior to receiving treatment.

Exclusion Criteria:

1. hypertensive patients with blood pressure exceed 160/100 mmHg;
2. a history of thrombosis,cerebrolvascular diseases, cancer, liver disease or liver dysfuction, hyperlipidemia, mental disorder, and severe infection;
3. having taken any pharmacological treatments affecting reproductive endocrine system;
4. having received acupuncture in the previous three months;
5. smoking more than 15 cigarettes per day;
6. having pacemakers, metal allergies or severe fear of acupuncture.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Doctor, Study Director — Guang'anmen Hospital
Locations (1):
- Beijing Hospital of Integrated Traditional Chinese and Western Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
to share data by publishing paper
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after the paper published around the year of 2020
Access Criteria: researchers who are interested in this area

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements on local newspapers and posters.Of the 116 individuals who were initially recruited for this trial, 56 were excluded,sixty participants were randomly assigned to acupuncture group (n = 30) or CPA/EE group (n = 30).
Groups:
- Tung's Acupuncture Group: The study took Tung's acupoints as main acupuncture points, which were Fuke, Huanchao, Tianhuang, Renhuang, as well as the traditional acupoints Guanyuan (CV4) and Zigong (EX-CA1).
- CPA/EE Group: CPA/EE were administered for 21 days consecutively. The patients then stopped taking the pills for seven days and, on the eighth day, continued to take the pills again for three menstrual cycles (28 day cycles).
Period: Overall Study
Arm/Group | Tung's Acupuncture Group | CPA/EE Group
Started | 30 | 30
Completed | 27 | 25
Not Completed | 3 | 5
Not completed — Pregnancy | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tung's Acupuncture | CPA/EE | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (4.18) | 28.53 (4.28) | 28.9 (4.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60
course of disease [Mean (Standard Deviation); unit: month] | 58.83 (54.04) | 36.10 (25.56) | 47.47 (43.45)

OUTCOME MEASURES:

1. Primary Outcome: Change in LH/FSH Ratio From Baseline to the End of Treatment
Description: the change in LH/FSH ratio, values after 12-week treatment minus the values at baseline
Time Frame: baseline and 12 weeks
Population: Sixty participants were randomly assigned to acupuncture group (n = 30) or CPA/EE group (n = 30). During the study period, one participant in the acupuncture group withdrew because of living far away from hospital, two participants in the CPA/EE group withdrew because of taking other medicine and health reason.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Tung's Acupuncture | CPA/EE
Number analyzed (Participants) | 29 | 28
ratio | -0.66 [-1.03 to -0.28] | -0.96 [-1.34 to -0.59]

2. Secondary Outcome: Change in LH/FSH Ratio From Baseline to the 24th Week
Description: the change in LH/FSH ratio, values at the 24th week minus the values at baseline
Time Frame: baseline to the 24th week
Population: During the long-term observation, three participants in the acupuncture group withdrew because of living far away from hospital, pregnancy and taking other medicine. Five participants in the CPA/EE group withdrew because of taking other medicine,pregnancy, losting contact and health reason.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Tung's Acupuncture | CPA/EE
Number analyzed (Participants) | 27 | 25
ratio | -0.39 [-0.77 to -0.01] | -0.44 [-0.85 to -0.24]

3. Secondary Outcome: Changes in LH From Baseline to the End of Treatment
Description: changes in luteinizing hormone(LH), values after 12-week treatment minus the values at baseline
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Tung's Acupuncture | CPA/EE
Number analyzed (Participants) | 29 | 28
mIU/mL | -3.92 [-5.74 to -2.09] | -5.66 [-7.84 to -3.48]

4. Secondary Outcome: Changes in FSH From Baseline to the End of Treatment
Description: changes in follicle-stimulating hormone (FSH), values after 12-week treatment minus the values at baseline
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Tung's Acupuncture | CPA/EE
Number analyzed (Participants) | 29 | 28
mIU/mL | -0.49 [-1.06 to 0.08] | -0.22 [-0.98 to 0.55]

5. Secondary Outcome: Changes in Body Mass Index (BMI) From Baseline to the End of Treatment
Description: the changes in BMI, values after 12-week treatment minus the values at baseline
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Tung's Acupuncture | CPA/EE
Number analyzed (Participants) | 29 | 28
kg/m^2 | -0.90 [-1.36 to -0.43] | -0.44 [-0.71 to -0.17]

6. Secondary Outcome: Changes in Total Testosterone (TT) From Baseline to the End of Treatment
Description: changes in total testosterone (TT) , values after 12-week treatment minus the values at baseline
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Tung's Acupuncture | CPA/EE
Number analyzed (Participants) | 29 | 28
nmol/L | -0.67 [-0.99 to -0.36] | -0.33 [-0.98 to -0.05]

7. Secondary Outcome: Changes in Ovarian Volume From Baseline to the End of Treatment
Description: changes in ovarian volume, values after 12-week treatment minus the values at baseline
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm^3
Arm/Group | Tung's Acupuncture | CPA/EE
Number analyzed (Participants) | 29 | 28
cm^3 | -1.70 [-3.68 to 0.28] | -1.03 [-2.84 to 0.77]

8. Secondary Outcome: Changes in Polycystic Ovary Number From Baseline to the End of Treatment
Description: the changes in polycystic ovary number, values after 12-week treatment minus the values at baseline
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: polycystic ovaries
Arm/Group | Tung's Acupuncture | CPA/EE
Number analyzed (Participants) | 29 | 28
polycystic ovaries | 0.00 [-1.00 to 0.00] | 0.00 [0.00 to 0.00]

9. Secondary Outcome: Changes in the Number of Bleeding Events From Baseline to the End of Treatment
Description: Changes in the number of bleeding events, values after 12-week treatment minus the values at baseline
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: bleeding events
Arm/Group | Tung's Acupuncture | CPA/EE
Number analyzed (Participants) | 29 | 28
bleeding events | 0.66 [0.33 to 0.98] | 1.21 [0.75 to 1.68]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: No serious adverse event happened, eleven adverse mild events were descriped in the data tables below.
Arm/Group | Tung's Acupuncture Group | CPA/EE Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 4/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tung's Acupuncture Group (N=30) | CPA/EE Group (N=30)
Transient bruises at the sites of needle insertion (Skin and subcutaneous tissue disorders) | 5 (9) | 0 (0)
post-treatment soreness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT02729545/Prot_SAP_000.pdf